CLINICAL TRIAL: NCT06757920
Title: The Use of Bronchoscopic Argon Plasma Coagulation in Endobronchial Carcinoid
Brief Title: "Bronchoscopic Argon Plasma Coagulation for Managing Endobronchial Carcinoid Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Sabry, Lecturer of chest diseases, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOB - Endobronchial Carcinoid
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Endobronchial Carcinoid
Keywords: Argon Plasma Coagulation; fiberoptic bronchoscopy; endobronchial carcinoid

STUDY DESIGN:
Intervention Model Description: Argon Plasma Coagulation via non contact probe for debulking and fulgration of the endobronchial carcinoid using fiberoptic bronchoscopy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- fiberoptic bronchoscopy in one group (Active Comparator): fiberoptic bronchoscopic argon plasma coagulation for palliation of endobronchial carc inoid
  Interventions: Procedure: bronchoscopic argon plasma coagulation

INTERVENTIONS:
Procedure: bronchoscopic argon plasma coagulation — Argon Plasma Cogulation for Debulking Endobronchial Carcinoid Using Fiberoptic Bronchoscopy

SUMMARY:
A small tube will go through the respiratory tract and a non contact cauterization will be done to the inside tumor

DETAILED DESCRIPTION:
fiberoptic bronchoscopy will go through the tracheobronchial tree and after localization of the tumor, argon plasma coagulation by initiation non contact electrocautery will be done to the tumor

ELIGIBILITY:
Inclusion Criteria:

1 - Cooperative patient with written informed consent. 2- Patients diagnosed with endobronchial carcinoid. 3- Patients fit for fiberoptic bronchoscopy. 4- Patients unwilling or unfit for surgery.

Exclusion Criteria:

1 -Poor karnofsky score. 2- Patients unwilling or unfit for bronchoscopy. 3- Extraluminal lesion. 4- Patients with pacemaker. 5- Forced expiratory volume 1 is less than one litre.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Dyspnea Borg Scale | one month
  scale from 0 to 4 according to the degree of improvement

CONTACTS AND LOCATIONS:
Overall Officials: mohamed sabry eltarhony, lecturer, Principal Investigator — Alexandria University
Locations (1):
- Chest Department -Faculty of Medicine, Alexandria, Azarita, Egypt

IPD SHARING:
Plan to Share IPD: No
because it is against the rules of the chest department

REFERENCES:
- See also: Successful treatment of endobronchial carcinoid using argon plasma coagulation — https://pubmed.ncbi.nlm.nih.gov/23168553/
- Available data/document: Study Protocol: msabry776@yahoo.com — https://pubmed.ncbi.nlm.nih.gov/17482984/ — very good